CLINICAL TRIAL: NCT04257968
Title: Long-term Vascular and Psychosocial Complications in Adolescent and Young Adult (AYA) Head and Neck Cancer Survivors.
Brief Title: Long Term Complications in Head and Neck Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL71550.091.19
Record Dates: First submitted 2019-10-17; First posted 2020-02-06 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2019-10

CONDITIONS: Head-and-neck Cancer
Keywords: Head and Neck Cancer; Radiotherapy; Complications; Vascular
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic intervention (Experimental): Complete diagnostic intervention
  Interventions: Diagnostic Test: Ultrasonography; Diagnostic Test: MRI; Diagnostic Test: Neuro Psychological Assessment Battery; Diagnostic Test: Questionaires

INTERVENTIONS:
Diagnostic Test: Ultrasonography — carotid ultrasonography (IMT and elastography)
Diagnostic Test: MRI — MRI of carotid artery and brain
Diagnostic Test: Neuro Psychological Assessment Battery — Hopkins Verbal Learning Test Digit Span WAIS-IV Stroop Color Word test Trail Making Test Brixton Spatial Anticipation Test Fluency letter (B-D-H) Fluency animal naming Symbol Digit Substitution WAIS-IV
Diagnostic Test: Questionaires — Cognitive Failures, Depression, Anxiety, Fatigue, Speech handicap, fear for recurrence, Quality of Life.

SUMMARY:
Problem:

With increasing numbers of cancer survivors, strategies to prevent long-term complications in cancer patients become more important. Adolescent and Young Adult (AYA) Head and Neck Cancer survivors treated with radiotheray (RT) are prone to long-term complications, especially vascular and psychosocial complications. Although several studies point to the importance of these long-term complications, structured survivorship care for AYA HNC survivors is still lacking.

Primary objective:

To investigate in AYA HNC survivors treated with unilateral RT at least 5 years before, the long-term vascular complications in terms of carotid wall changes (ultrasonography, MRI), cerebral vascular complications ((silent)brain infarctions, white matter lesions) and Cardiovascular Risk Management profile.

Secondary objective:

To investigate in AYA HNC survivors treated with unilateral RT at least 5 years before, the long-term psychosocial complications (subjective memory complaints, Depression, Anxiety, Fatigue, Speach handicap, Anxiety for recurrence, Quality of Life, objective cognitive failure)

Study design Prospective cohort study.

Patient population AYA HNC survivors ≥ 5 years after unilateral RT, either alone or in combination with surgery and/or chemotherapy.

Controls The ultrasonography (Intima Media Thickness, elastography) and MRI measurements of the irradiated carotid wall will be compared to the non-irradiated carotid wall. Cognitive performance will be compared to normative data. The cognitive performances of the right hemisphere tests will be compared to the cognitive performances of the left hemisphere tests. The frequency of silent brain infarcts and vascular white matter lesions of the irradiated vascular territory will be compared with the non-irradiated territory.

Intervention Structured survivorship care ≥ 5 years after RT conform the Personalized Cancer Survivorship Care Model of the Radboudumc Expertisecenter of late effects after cancer, complemented with carotid ultrasonography (IMT and elastography), MRI of the carotid arteries and brain), neuropsychological assessment battery and self-reported questionnaires concerning depression, fatigue, QoL, positive health and employment status.

ELIGIBILITY:
Inclusion Criteria:

* HNC patient treated with unilateral RT at age 18-40 years 5-10 years before
* Informed Consent

Exclusion Criteria:

* Contra indication MRI
* Able to communicate in Dutch language

Ages: 23 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-01-22 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Intima Media Thickness (mm) | 5-10 years after radiotherapy
  Intima Media thickness in mm on ultrasonography in the irradiated versus the non irradiated carotid artery
Carotid wall elastography | 5-10 years after radiotherapy
  Carotid wall elastography on ultrasonography in the irradiated versus the non-irradiated artery:
  distense coëfficiënt, pulse wave velocity (PWV) (during diastole and systole) and shear wave velocity (SWV) (2-8 moments during heartbeat)
Carotid wall thickness on MRI (mm) | 5-10 years after radiotherapy
  Carotid wall thickness in mm on MRI in the irradiated versus the non-irradiated artery
Radiological characteristics of carotid wall changes on MRI | 5-10 years after radiotherapy
  Radiological characteristics of carotid wall changes on MRI of the irradiated versus the non-irradiated artery: intensity on T1/T2/FLAIR/Proton Density.
Pack Years smoking | 5-10 years after radiotherapy
  Pack Years smoking
Hypertension | 5-10 years after radiotherapy
  Definition: Systolic Bloodpressure > 140 mmHg or taking antihypertensive medication
Cardiovascular risk management: Body Mass Index | 5-10 years after radiotherapy
  weight and height will be combined to report BMI in kg/m^2
White matter hyperintensities on MRI | 5-10 years after radiotherapy
  Volume of white matter hyperintensities on FLAIR in ml
Number of brain infarctions on MRI | 5-10 years after radiotherapy
  Number of brain infarctions assessed on MRI

SECONDARY OUTCOMES:
Subjective Memory Complaints | 5-10 years after radiotherapy
  Assessed by Cognitive Failure Questionairre:
  a questionairre about failures in perception, attention, memory, and motor function.
  29 items Total score Range 0-100
Cognitive function | 5-10 years after radiotherapy
  Cognitive function per cognitive domain:
  Available normative data will be used to convert the patients results on the neuropsychological tests into standardized T scores (mean, SD), adjusted for age, sex and education.
Hospital Anxiety and Depression Scale (HADS). | 5-10 years after radiotherapy
  Hospital Anxiety and Depression Scale (HADS). The total scores range is 0-21 for both depression and anxiety scores. A higher score indicates a worse depression and anxiety.
  14 items Score depression: Range 0-21 Score Anxiety: Range 0-21 Total score: Range 0-42
Fatigue severity | 5-10 years after radiotherapy
  Fatigue severity was assessed using the Checklist Individual Strength (CIS20R), a 20-item questionnaire that takes around five to ten minutes to fill out. Each question has a statement to be scored on a 7-point Likert scale ranging between 'yes, this is true' to 'no, this is not true'. The total score is calculated as the sum of the responses to the different statements. The maximum CIS20R score is 140, with a score of 76/140 or higher indicating that the patient is at risk for prolonged absence at work. The scale is subdivided in four dimensions of fatigue being fatigue severity (8 items, max. score 56), concentration problems (5 items, max. score 35), reduced motivation (4 items, max. score 28) and activity (3 items, max. score 21).
  Total score: Range 20-140
Speech Handicap Index (SHI) | 5-10 years after radiotherapy
  Assessed by Speech Handicap Index:
  a questionairre assessing self perceived speech function. 30 items A total SHI can be calculated ranging from 0-120, with higher scores indicating more speech problems and with a cutoff value of 6 being able to identify patients with speech problems in daily life.
Brief symptoms Inventory (BSI) | 5-10 years after radiotherapy
  Assessed by Brief Symptom Inventory measure Brief Symptom Inventory (BSI) measure consists of 18 emotional distress items that are rated on a 5 point Likert scale and yield a Global Severity Index as well as Symptom Dimensions (Somatization, Depression, Anxiety.
  Total score: Range 0-72
Fear of recurrence | 5-10 years after radiotherapy
  Assessed by the Cancer Worry Scale (CWS):
  self reported 8-item scale, measuring worry about the risk of cancer recurrence and its impact on daily functioning. Total score ranges from 8 to 32. Higher scores indicate higher FCR. A cutoff score of 13 vs 14 (low FCR 13 or lower; high FCR 14 or more) has been established to differentiate between those with normal FCR from those with bothersome levels of FCR. This cutoff had been validated relative to the Fear of Cancer Recurrence Inventory cutoff score, which is a validated maesure.
Cancer specific distress | 5-10 years after radiotherapy
  Assessed by Impact of Event Scale-Revised, which is a 22-items scale and includes subscales of intrusion, sleep disturbance, hyperarousal, avoidance and numbing. Items are scored on a 5-point scale, ranging from 0 (not at all) to 4 (extremely).
Quality of Life | 5-10 years after radiotherapy
  Assessed using the EORTC-QLQ-C30 questionairre consisting of 30 items. Total score: Range 0-100

CONTACTS AND LOCATIONS:
Overall Officials: Hans Kaanders, MD, PhD, Prof, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboudumc, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pruijssen JT, Wilbers J, Meijer FJA, Pegge SAH, Loonen JJ, de Korte CL, Kaanders JHAM, Hansen HHG. Assessing radiation-induced carotid vasculopathy using ultrasound after unilateral irradiation: a cross-sectional study. Radiat Oncol. 2022 Jul 23;17(1):130. doi: 10.1186/s13014-022-02101-7. PMID 35871069
- [Derived] Pruijssen JT, Wenmakers A, Kessels RPC, Piai V, Meijer FJA, Pegge SAH, Loonen JJ, Tuladhar AM, Hansen HHG, Kaanders JHAM, Wilbers J. Long-term cognitive, psychosocial, and neurovascular complications of unilateral head and neck irradiation in young to middle-aged adults. BMC Cancer. 2022 Mar 5;22(1):244. doi: 10.1186/s12885-022-09295-9. PMID 35248013